CLINICAL TRIAL: NCT05310890
Title: Long Term Prospective Study of Tai Chi Intervention to Prevent MCI From Conversion to Dementia
Acronym: TIME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Zhangjiagang Aoyang Hospital of Jiangsu Province (Unknown)
Responsible Party: Principal Investigator, Shengdi Chen, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TIME study
Record Dates: First submitted 2022-03-17; First posted 2022-04-05 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Tai Chi
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai chi training plus group activity (Experimental): Tai chi training: a teacher will give two 60-min lessons per week. Participants will play Tai Chi in the lessons, following teacher's instruction.
  Group activity: a organizer will lead the subjects to participate in group activities, once per quarter.
  Interventions: Behavioral: Tai chi training; Behavioral: Group activity
- Only group activity (Other): Group activity: a organizer will lead the subjects to participate in group activities, once per quarter.
  Interventions: Behavioral: Group activity

INTERVENTIONS:
Behavioral: Tai chi training — Tai chi, also called tai chi chuan, is an ancient Chinese form of exercise originally created as a fighting art. It is a kind of gentle physical exercise and stretching, which involves a series of movements performed in a slow, focused manner and accompanied by deep breathing.
  Arms: Tai chi training plus group activity
Behavioral: Group activity — A organizer will lead the subjects to participate in group activities once a quarter. In group activities, there will be popular science lectures and interactive games.

SUMMARY:
This study evaluates the effects of 3 years-Tai Chi exercise intervention on cognitive function in MCI patients and to clarify whether the intervention can prevent MCI from conversion to dementia. Patients will be randomized into the Tai chi training group and the control group.

DETAILED DESCRIPTION:
Dementia is a syndrome of impairments of cortical functions caused by brain diseases. More than 55 million people worldwide are currently living with dementia, with nearly 10 million new cases each year. Alzheimer's disease is the most common form of dementia and may account for 60-70% of patients with dementia. Mild cognitive impairment (MCI) is an intermediate state between normal cognitive aging and dementia. About 10% to 15% of patients with MCI progress to dementia each year. Therefore, it is crucial to find intervention strategies to prevent the progression of MCI to dementia. However, drug interventions are currently ineffective in the prevention of dementia. Based on the synaptic plasticity, more and more studies focus on non-drug interventions. Our research group previously found 6-months non-drug interventions (cognitive training, exercise therapy) can effectively delay cognitive decline in the elderly, providing a new strategy for the improvement of cognition in the elderly. Therefore, this project plans to conduct a multi-site, randomized, parallel-controlled clinical trial to examine the effect of 3 years-Tai Chi exercise intervention on cognitive function in MCI patients and to clarify whether the intervention can prevent MCI from conversion to dementia.

ELIGIBILITY:
Inclusion Criteria

1. Male and female participants aged 55 to 85 years (inclusive) at the time of screening
2. Willing and able to give informed consent by GCP and local guidance.
3. Meets the National Institute on Aging of the National Institutes of Health and Alzheimer's Association (NIA-AA) diagnostic criteria for "Mild Cognitive Impairment Due to Alzheimer's Disease" (2011); does not meet the American Psychiatric Association's diagnostic criteria Diagnostic and Statistical Manual of Mental Disorders, Revised IV (DSM-IV-R) diagnostic criteria for dementia;
4. Main complaint of memory loss, 24≤MMSE and/or 17≤MOCA<26 points, with one or more cognitive domains impairments;
5. CDR global score of 0.5, with memory box score ≥0.5
6. Functional activities questionnaire (FAQ) <5
7. Hachinski ischemia score ≤4;
8. Have the physical, cognitive, listening, speech, literacy and language skills necessary to participate in all tests;
9. Capable of performing MR
10. Allowed and Prohibited concomitant and treatments.

During the clinical study, the following drugs are prohibited:

Acetylcholinesterase inhibitors, N-methyl-D-aspartate (NMDA) antagonists (eg, memantine, amantadine, ketamine, and dextromethorphan), adrenal corticosteroids, central nervous system stimulants, traditional Chinese medicine and various medicines that can improve memory or cognition;

During the clinical study, the following drugs cannot be added:

Antipsychotics, antidepressants, sedative-hypnotics for sleep (zopiclone, alprazolam, estazolam can be used temporarily if necessary) For long-term use of the above drugs, the dose should be kept as stable as possible during the study.

Exclusion Criteria

1. Cognitive impairment caused by other reasons (for example) cerebrovascular disease, central nervous system infection, Creutzfeldt-Jakob disease, Huntington's disease, Parkinson's disease, dementia with Lewy bodies, trauma, other physical and chemical factors (drugs, alcohol, CO, etc.), important physical diseases (hepatic encephalopathy, pulmonary encephalopathy, etc.), brain tumor, endocrine diseases (thyroid disease, parathyroid disease), and vitamin deficiency or any other cause of dementia;
2. Abnormal folate, thyroid, and/or vitamin B12 values that cannot be corrected before baseline visit.
3. Major structural brain disease as judged by central MRI Diagnostic Imaging Review Team (eg, ischemic infarcts, subdural hematoma, hemorrhage, hydrocephalus, brain tumors, multiple subcortical ischemic lesions. or a single lesion in a critical region [eg, thalamus]). Mild white matter changes without clinical significance and no more than 2 lacunar infarcts are permitted.
4. Mental illness determined by Diagnostic and Statistical Manual of Mental Disorders (DSM) V criteria, that is unstable within 12 months, or would interfere with study assessments, including schizophrenia or other psychotic disorders, bipolar disorder, severe depression, or delirium.
5. DSM V diagnosis of alcohol or other substance abuse dependence within the last 12 months.
6. History or current diagnosis of significant cardiac arrhythmias, myocardial infarction, transient ischemic attack, or cerebrovascular accident, uncompensated congestive heart failure New York Heart Association class III and IV.
7. Major medical illness or unstable medical condition within 6 months of screening that in the opinion of the investigator may interfere with the participant's ability to comply with study procedures and abide by study restrictions, or with the ability to interpret safety data, including any physical disability (eg. blindness. deafness, non-cognitive related speech impairment, sensory or motor dysfunction) that would prevent completion of study procedures or assessments.
8. Cancer except:

   1. History of any cancer that has been in remission (no evidence of recurrence) for > 3 years from the screening
   2. Participants with basal cell or stage I squamous cell carcinoma of the skin, stable untreated cancer as prostate or meningioma.
9. Exercise regularly within 6 months prior to screening.
10. Participants are excluded if they

    1. have participated in any other clinical study within 4 weeks prior to screening visit
    2. have participated in another Tai chi clinical study at any time
    3. plan to take part in another clinical study during this study.
11. Geriatric Depression Scale-15(GDS-15) total score > 7 at screening
12. The researcher estimates that the subject's compliance is poor, and it is believed that the subject is unlikely to complete the study.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of MCI converted to Alzheimer's disease. | 36 months
  The 3-year incidence of AD in each group will be compared.
The global cognitive function of MCI patients. | 18 months and 36 months
  11-item Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog 11) will be used to assess the global cognitive performance of MCI patients. The total score of ADAS-cog/11 is 0-70, with higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Memory | 18 months and 36 months
  Memory will be assessed using the Auditory verbal learning test-Huashan version (AVLT-H).
Attention | 18 months and 36 months
  Attention will be evaluated by Trial Making Test (TMT).
Executive function | 18 months and 36 months
  Executive function will be evaluated by the Stroop task.
Language | 18 months and 36 months
  Language will be assessed by Boston naming test (30-item version), and Verbal Fluency.
Working memory test | 18 months and 36 months
  Working memory test will be assessed by Number Span Forward and Backward.
Visual spatial ability | 18 months and 36 months
  Visual spatial ability will be assessed by Clock Drawing Test.
Change from baseline in MMSE score | 18 months and 36 months
  Change from baseline in Mini Mental State Examination (MMSE) score. The total score of MMSE is 0-30, with higher scores mean a better outcome.
Change from baseline in MoCA score | 18 months and 36 months
  Change from baseline in Montreal Cognitive Assessment (MoCA) score. The total score of MoCA is 0-30, with higher scores mean a better outcome.
Change from baseline in CDR score | 18 months and 36 months
  Change from baseline in Clinical Dementia Rating (CDR) Scale score.
Activities of daily living | 18 months and 36 months
  Activities of daily living will be assessed by functional activities questionnaire (FAQ). The total score of FAQ is 0-30, with higher scores mean a worse outcome.
Anxiety | 18 months and 36 months
  Anxiety will be assessed by Hamilton Anxiety Rating Scale (HAMA).The total score of HAMA is 0-56, with higher scores mean a worse outcome.
Depression | 18 months and 36 months
  Depression will be assessed by Hamilton Depression Rating Scale (HAMD).
Sleep | 18 months and 36 months
  Sleep will be assessed by Pittsburgh Sleep Quality Index (PSQI).The total score of PSQI is 0-21, with higher scores mean a worse outcome.
Brain activity | 36 months
  Detecting changes associated with blood flow by fMRI.
Neurodegeneration in brain structures | 36 months
  Brain atrophy will be assessed by Magnetic Resonance Volume Imaging.
Gut microbiota | 18 months and 36 months
  Gut microbiota will be assessed by 16S rRNA sequencing.
Blood biomarkers | 18 months and 36 months
  Inflammatory factors (FGF basic、Eotaxin、G-CSF、GM-CSF、IFN-γ、IL-1β、IL-1ra、IL-2、IL-4、IL-5、IL-6、IL-7、IL-8、IL-9、IL-10、IL-12 (p70)、IL-13、IL-15、IL-17、IP-10、MCP-1 (MCAF)、MIP-1α、MIP-1β、PDGF-BB、RANTES、TNF-α、VEGF) will be measured by Bio-Plex Human Cytokine Assays.

IPD SHARING:
Plan to Share IPD: No